CLINICAL TRIAL: NCT04586595
Title: A Randomised Pilot Study of a Pharmacist-led Retrospective Review of Prescribing by General Practitioners in Training (REVISiT) Intervention
Brief Title: A Randomised Pilot Study of the REVISiT Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19007
Record Dates: First submitted 2020-08-06; First posted 2020-10-14 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Patient Safety; Inappropriate Prescribing; Medication Errors
Keywords: General practice; Pharmacist role; GP training; Educational interventions

STUDY DESIGN:
Intervention Model Description: Parallel two-arm randomised pilot study
Who Masked: Outcomes Assessor
Masking Description: Researchers responsible for analysis of error rate and rate of suboptimal prescribing will not know which arm the results have come from
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): GP trainees in this arm will receive the REVISiT intervention which will involve having their prescribing reviewed and feedback provided, at two time points (approximately 100 prescriptions at each time point) separated by approximately a 3-month time period.
  Interventions: Other: REVISiT intervention
- Control arm (No Intervention): GP trainees in this arm will continue with training as usual and will have their prescribing (approximately 200 prescriptions) reviewed once but representing two time points - separated by an approximate 3-month time period. Feedback will occur at one time point, to cover the review for the 200 prescriptions.

INTERVENTIONS:
Other: REVISiT intervention — REVISiT is a pharmacist-led retrospective review of prescribing followed by a feedback meeting to discuss the review findings.
  Arms: Intervention arm

SUMMARY:
In 2012, the General Medical Council (GMC) funded PRACtICe (PRevalence And Causes of prescrIbing errors in general practiCe) study, reported that 1 in 20 prescriptions in general practice were found to have a prescribing or monitoring error. The PRACtICe study also proposed some strategies to consider to improve prescribing safety.

Further to the PRACtICe study, in line with recommendation from the Medical Research Council (MRC) for developing complex interventions, we conducted a series of focus groups with health care professionals and members of the public to identify possible ways to improve the prescribing education provided for general practitioner (GP) trainees - a group that was identified as likely to benefit from additional education and training in prescribing safety. These focus group discussions identified a pharmacist-led review of the prescribing done by GP trainees, together with feedback, as a promising potential intervention. This intervention, named REVISiT, was piloted with ten trainees and their trainers in the East Midlands. The error rate for the trainees was recorded as 9%. Interviews with the trainees and trainers undertaken following the intervention highlighted that REVISiT was positively received. Some GPs gave examples of how their prescribing practice had changed following the intervention.

After this pilot study, we conducted another study involving interviews, focus groups and a stakeholder event with key stakeholders (practice, policy, legal and members of the public) to explore the next steps for REVISiT. Whilst some participants proposed that REVISiT be immediately implemented with minor modifications, others pointed to the need to establish the impact of the intervention more broadly (including its impact in areas other than education and training). Additionally, they highlighted the importance of establishing its effectiveness in order to support making a substantial case for future allocation of resources. Conducting a randomised controlled trial (RCT) would help establish the effectiveness of the REVISIT intervention and its impact on areas of professional practice that may impact prescribing safety. However, before we can do this, there are components of the REVISiT intervention and RCT process that we need to further explore, test and refine in order for it to be employed on a wider basis. This pilot study of the REVISiT intervention is being undertaken to do this further exploration, testing and refining.

DETAILED DESCRIPTION:
Prescribing medication is integral to the role of a general practitioner (GP). Figures from 2017 show that an estimated 1,105.8 million prescription items were dispensed in England alone. However, in practice, sometimes prescribing errors occur and these have the potential to cause significant morbidity and mortality. The General Medical Council (GMC) funded PRACtICe study which set out to determine the prevalence and nature of prescribing and monitoring errors in general practices in England identified prescribing errors in around one in twenty prescriptions. The study also put forward explanations as to why some of the errors may have occurred and offered recommendations for strategies and areas of focus that could potentially be explored to improve prescribing. One of these areas highlighted for consideration was providing further support for prescribing, specifically for GPs in training. The study found that, as a group, GPs in training did not necessarily receive training in prescribing that was comprehensive and structured. GPs in training also reported feeling unprepared for managing patients with complex and long term health needs.

Further to the PRACtICe study, in line with recommendation from the Medical Research Council (MRC) for developing complex interventions4, a series of focus groups5 were convened with health care professionals and members of the public to explore in more details which ideas proposed as part of the PRACtICe study should be considered for further development. The results further highlighted the desire for GPs in training to receive further educational input in the area of prescribing practice and safety. Furthermore, an educational intervention considered that could potentially meet this training need, was an individualised, pharmacist-led retrospective review of GPs in training prescribing practice (REVISiT intervention).

Following on from the focus group study, a small pilot study was conducted in the East Midlands to explore the feasibility of using the REVISiT intervention in general practice.6 The REVISiT intervention itself started with a primary care pharmacist undertaking a retrospective review of approximately 100 consecutive prescription items prescribed by ten GPs in training (in total 1028 prescriptions were reviewed). This was then followed by each GP in training, and their trainer receiving individualised feedback in a form of a report. The report presented the GP with areas where errors were identified and examples of 'good prescribing'. The impact of the intervention on prescribing and the experience of participating in the pilot study was assessed qualitatively. For this, GPs in training and their trainers participated in two interviews, one was conducted within a month of receiving feedback and the second one within 3-months of receiving feedback. Results from this pilot study reported an error rate of 9%, which was higher than the 5% error rate recorded in the GMC PRACtICe study. Furthermore, the pharmacist review identified a high rate of 'suboptimal' prescribing (35% of prescriptions) which identified further areas where GPs in training could improve on their prescribing. The qualitative narratives revealed that the REVISiT intervention was positively received by GPs and was deemed a unique training opportunity to receive individualised feedback on prescribing skills and knowledge that had potential to improve their prescribing and subsequently patient safety. GPs in training gave examples of where their prescribing had changed as a result of the REVISiT intervention and some communicated their intention to change, or implement a prescribing behaviour when the next opportunity arose.

After the pilot study, we conducted a qualitative study involving interviews, focus groups and a stakeholder event with key stakeholders (practice, policy, legal and members of the public) to explore whether the REVISiT intervention, in its current or modified form, should be considered for wide spread adoption into GP training and general practice or whether an evaluation study to establish the effectiveness and cost-effectiveness of the intervention was first warranted. Some participants expressed their disbelief that an intervention such as REVISiT was not already in routine use in general practice. They mainly felt that with some modifications the intervention would be fit to recommend for use. On the contrary, some suggested that more robust evidence, generated from conducting a definitive randomised controlled trial, would be needed before directing already limited resources towards an intervention in its early stages of development and use such as REVISiT.

However, before we are able to conduct a definitive randomised controlled trial of the REVISiT intervention to assess its effectiveness in improving prescribing of GPs in training (increase in the proportion of prescriptions prescribed correctly / reduction of observed prescribing errors) and the cost-effectiveness, there are components of the intervention itself and the trial process that need to be further explored, tested and refined. This step is important because there is evidence in the literature pointing to the 'failure' of some interventions arising due to poor intervention and study design and description.4

ELIGIBILITY:
Inclusion Criteria:

* Participants who are able and willing to give written informed consent and are either:
* GPs in their final year of training who have received approval/permission from their GP trainer to participate in the study or;
* GP trainers with a trainee who has consented to take part in the pilot study or;
* Primary care pharmacists (employed by the practice, the primary care network (PCN) or the clinical commissioning group (CCG) in which the GP in training works) with ideally, at least 6-months experience of working in GP practices or;
* Pharmacists specially trained to deliver the REVISiT intervention and trained on good clinical practice (GCP) in research

Exclusion Criteria:

* Participants not able or willing to give written informed consent
* GP trainees with significant participation in other studies that could impact / could be impacted by their taking part in this randomised pilot study
* GP trainees who do not have the support of their trainer to participate in the study
* GP trainers who do not wish for their trainee to be involved with the study
* Pharmacists who do not have the required experience (ideally at least 6-month) of working in general practice in England
* Pharmacists who are not trained in delivering the REVISiT intervention or on GCP as part of this study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Change in the prevalence and types of prescribing errors | The first review of prescribing corresponds to a time of no more than 4 weeks post baseline. The comparative review of prescribing corresponds to a time of no more than 20 weeks post baseline
  Prescribing errors will be identified following a pharmacist-led retrospective review of prescribing done by GP trainees to assess the impact of the REVISIT intervention on the types and numbers of prescribing errors

SECONDARY OUTCOMES:
Change in the prevalence and types of suboptimal prescribing | The first review of prescribing corresponds to a time of no more than 4 weeks post baseline. The comparative review of prescribing corresponds to a time of no more than 20 weeks post baseline
  Suboptimal prescribing will be identified following a pharmacist-led retrospective review of prescribing done by GP trainees to assess the impact of the REVISIT intervention on the types and numbers of suboptimal prescribing observed
Participant recruitment and attrition | Study completion
  Will include the number of participants recruited and completing the study as per study group allocation (where possible, reasons for declining participation or withdrawal from the study will be recorded)
Interrater reliability between review pharmacists | The first review of prescribing corresponds to a time of no more than 4 weeks post baseline. The comparative review of prescribing corresponds to a time of no more than 20 weeks post baseline
  Each review pharmacist will have 10% of their prescribing review, coded by a second pharmacist to provide an assessment of interrater reliability with regards to the prescribing errors and suboptimal prescribing identified
Sample size estimation for the definitive randomised controlled trial | Study completion - estimated to be one year after the commencement of the study
  Data generated from the randomised pilot study will be used to estimate a sample size for the definitive randomised controlled trial
Experiences of participants in relation to the randomised controlled trial | This will take place at a time no longer than 24 weeks post baseline
  Participants will be involved in a semi-structured interview to explore their experiences of participating in the randomised controlled trial including allocation and adherence to study treatment groups; and to explore what modifications, if any, may enhance the acceptability and success of conducting a future definitive randomised controlled trial of the REVISiT intervention in general practice
Experiences of participants in relation to the REVISiT intervention | This will take place at a time no longer than 24 weeks post baseline
  Participants will be involved in a semi-structured interview to explore their experiences of the REVISiT intervention including (where relevant) the - pharmacist training, database, REVISiT case-law for guiding the review process, mechanisms of action (e.g. whether feedback increases capability and motivation) and the impact of the prescribing review on current and future prescribing practice.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Knox, MBChB, Principal Investigator — University of Nottingham; Nde-Eshimuni M Salema, PhD, Study Director — University of Nottingham; Anthony J Avery, DM, Study Director — University of Nottingham; Darren Ashcroft, PhD, Study Director — University of Manchester; Chris Armitage, PhD, Study Director — University of Manchester; Brian Bell, PhD, Study Director — University of Nottingham; Glen Swanwick, Study Director — Patient and Public Involvement; Jeanne-Anna Charly, Study Director — Patient and Public Involvement; Gill Gookey, Study Director — Clinical Commissioning Group collaborators; Mindy Bassi, Study Director — Clinical Commissioning Group collaborators; Richard Williams, BA, Study Director — University of Manchester
Locations (4):
- United Kingdom (4):
  - NHS Derbyshire, Derby, Derbyshire
  - NHS Lincolnshire, Lincoln, Lincolnshire
  - NHS Nottingham, Nottingham, Nottinghamshire
  - NHS Dorset CCG, Dorchester

IPD SHARING:
Plan to Share IPD: No
Only named researchers in the study team will have access to individual participant data - and only if necessary for the completion of the study

REFERENCES:
- [Background] Duerden M, Millson D, Avery A and Smart S. The quality of GP prescribing: An Inquiry into the Quality of General Practice in England. 2011.
- [Background] Avery T, Barber N, Ghaleb M, Franklin BD, Armstrong S, Crowe S, Dhillon S, Freyer A, Howard R, Pezzolesi C, Serumaga B, Swanwick G and Talabi O. Investigating the prevalence and causes of prescribing errors in general practice: The PRACtICe Study (PRevalence And Causes of prescrIbing errors in general practiCe). London: A report for the GMC; 2012.
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Marsden K, Avery T, Knox R, Gookey G, Salema N and Bassi M. Focus group study to explore ideas on potential interventions for reducing prescribing errors in general practice. Pharmacoepidemiology and Drug Safety. 2013; 22:681
- [Background] Knox R, Gookey G, Salema N, Marsden K, Swanwick G, Bassi M, Silcock N, Bell B, Mehta R, Rodgers S, Coulton A and Avery T, 2017. Retrospective review of prescriptions issued by GPs in training - a pilot study. Pharmacoepidemiology and Drug Safety. 2017; 26: 3-20.
- [Background] Knox R, Salema N, Gookey G, Marsden K, Bell B, Mehta R, Roders R, McCartney K and Avery T. REVISIT, the next stage: developing plans for wider application of a retrospective review of prescribing of GPs in training. British Journal of General Practice. 2018; 68 (suppl 1): bjgp18X697337.
- [Background] Carver CS, Scheier MF. Control theory: a useful conceptual framework for personality-social, clinical, and health psychology. Psychol Bull. 1982 Jul;92(1):111-35. No abstract available. PMID 7134324